CLINICAL TRIAL: NCT01555619
Title: Quadripolar Pacing Post Approval Study
Acronym: Quad PAS
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 60030283
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure
Keywords: Left heart pacing lead; Cardiac resynchronization therapy (CRT); Heart Failure; Quadripolar pacing
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- CRT-D System: St. Jude Medical (SJM) Promote® Q/Promote® Quadra/Unify Quadra™ CRT-D system.
  Interventions: Device: CRT-D System

INTERVENTIONS:
Device: CRT-D System — Implantation of a CRT-D System
  Other Names: CRT-D and LV pacing lead

SUMMARY:
The purpose of this post-approval study is to evaluate the acute and chronic performance of a Quadripolar CRT-D device system in a patient population indicated for cardiac resynchronization therapy (CRT).

DETAILED DESCRIPTION:
Quad PAS is a multi-center, post-approval study. Patients who meet inclusion/exclusion criteria will have an attempted implant of a Quadripolar CRT-D device system (device and left ventricular (LV) lead). Patients who have an unsuccessful implant will be followed for 30 days for any adverse events and then withdrawn from the study, or may have an implant reattempted if the physician chooses to do so. Patients enrolled in the study will be followed at 6 months, and every 6 months thereafter, for 60 months of follow up (5 years). After patients complete 60 months of follow-up, their participation in the study will be terminated.

ELIGIBILITY:
Inclusion Criteria:

1. Approved indication per current American College of Cardiology/American Heart Association/Heart Rhythm Society guidelines for implantation of a CRT-D system for treatment of heart failure or life threatening ventricular tachyarrhythmia(s).
2. Participated in the Promote® Q CRT-D and Quartet™ Left Ventricular Heart Lead Study (Investigational Device Exemption (IDE) study), or are receiving a new Quadripolar CRT-D device system implant or are undergoing an upgrade from an existing implantable cardioverter-defibrillator or pacemaker implant with no prior LV lead placement.
3. Have the ability to provide informed consent for study participation and be willing and able to comply with the prescribed follow-up tests and schedule of evaluations

Exclusion Criteria:

1. Have a hypersensitivity to a single 1.0mg dose of dexamethasone sodium phosphate
2. Have a life expectancy of less than 5 years due to any condition
3. Be less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for CRT.
Sampling Method: Non-Probability Sample
Enrollment: 1971 (Actual)
Dates: Start 2012-02-15 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Complication free survival rate related to the CRT-D system | 5 years
  Complication free survival rate through 5 years for complications related to the CRT-D system
Complication free survival rate related to the LV lead | 5 years
  Complication free survival rate at 5 years for complications related to the LV lead
Mean programmed LV lead pacing capture threshold | 5 years
  Mean programmed LV lead pacing capture threshold at 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Corbisiero, MD, Study Chair — Deborah Heart and Lung Center
Locations (71):
- United States (71):
  - Cardiology, P.C., Birmingham, Alabama
  - Heart Center Research, LLC/Research Center, Huntsville, Alabama
  - Southeastern Cardiology Consultants PC, Montgomery, Alabama
  - Arizona Arrhythmia Research Center, Phoenix, Arizona
  - Washington Regional Medical Center, Fayetteville, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Comprehensive Cardiovascular, Bakersfield, California
  - Scripps Green Hospital, La Jolla, California
  - USC Unversity Hospital, Los Angeles, California
  - Fogarty Institute, Mountain View, California
  - Premier Cardiology, Inc., Newport Beach, California
  - Cardiac Rhythm Specialists, Inc., Northridge, California
  - St. Joseph Heritage Medical Group, Orange, California
  - Regional Cardiology Associates, Sacramento, California
  - St. Joseph's Medical Center, Stockton, California
  - Cardiology Associates Medical Group, Inc., Ventura, California
  - Florida Electrophysiology Associates, Atlantis, Florida
  - Yoel R. Vivas, MD, Boynton Beach, Florida
  - Jorge Diaz, Lake Mary, Florida
  - Naples Heart Rhythm Specialists, Naples, Florida
  - Munroe Regional Medical Center, Ocala, Florida
  - Florida Heart Rhythm Specialists, LLC, Plantation, Florida
  - Northside Hospital, St. Petersburg, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Piedmont Heart Institue, Atlanta, Georgia
  - HeartCare Midwest, Peoria, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Northwest Indiana CardiovascularPhysicians, P.C., Munster, Indiana
  - Unity Point Clinic, Cedar Rapids, Iowa
  - Central Baptist Hospital, Lexington, Kentucky
  - Northeast Cardiology Associates, Bangor, Maine
  - MedStar Health Research Institute, Baltimore, Maryland
  - Shady Grove Adventist Hospital, Rockville, Maryland
  - Lahey Clinic, Burlington, Massachusetts
  - Sinai Grace Hospital, Detroit, Michigan
  - Thoracic Cardio Healthcare Foundation, Lansing, Michigan
  - Missouri Baptist Medical Center, St Louis, Missouri
  - The International Heart Institute of Montana, Missoula, Montana
  - Heart Consultants P.C., Omaha, Nebraska
  - Cardiovascular Consultants of Nevada, Las Vegas, Nevada
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Cardiovascular Associates of the Delaware Valley, Haddon Heights, New Jersey
  - Presbyterian Heart Group, Albuquerque, New Mexico
  - Albany Medical College at Albany Medical Center, Albany, New York
  - Stonybrook University Medical Center, Stony Brook, New York
  - Buffalo Cardiology & Pulmonary Association, Williamsville, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Caromount Heart, Gastonia, North Carolina
  - Sanford Research, Fargo, North Dakota
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - EMH Regional Medical Center, Elyria, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Bryn Mawr Medical Specialists Associates, Bryn Mawr, Pennsylvania
  - Saint Vincent Consultants in Cardiovascular Diseases, Erie, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pee Dee Cardiology Associates, PA, Florence, South Carolina
  - Cardiology Consultants, Johnson City, Tennessee
  - Cardiovascular Associates, PC, Kingsport, Tennessee
  - Arrythmia Consultants, P.C., Memphis, Tennessee
  - St. Thomas Hospital, Nashville, Tennessee
  - HeartPlace, Bedford, Texas
  - Cardiology Associatesof Corpus Christi, Corpus Christi, Texas
  - Houston Arrhythmia Associates, Houston, Texas
  - Medicine School of University Health Care, Salt Lake City, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Harrisonburg Medical Associations, Inc., Harrisonburg, Virginia
  - Virginia Cardiovascular Specialists, Richmond, Virginia
  - Heart Clinics Northwest, Spokane, Washington
  - Morgantown Internal Medicine Group, Inc., Morgantown, West Virginia
  - Aspirius Heart and Vascular Institute, Research and Education, Wausau, Wisconsin

IPD SHARING:
Plan to Share IPD: No